CLINICAL TRIAL: NCT00849147
Title: A Multi-Center, Phase II Trial of Nonmyeloablative Conditioning (NST) and Transplantation of Partially HLA-Mismatched Bone Marrow From Related Donors for Patients With Hematologic Malignancies (BMT CTN #0603)
Brief Title: Bone Marrow Transplant From Partially Matched Donors and Nonmyeloablative Conditioning for Blood Cancers (BMT CTN 0603)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN0603; U01HL069294 (NIH); 5U24CA076518 (NIH)
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse
Keywords: Acute Lymphoblastic Leukemia/Lymphoma; Acute Myelogenous Leukemia; Mantel-Cell Lymphoma; Hematopoietic Transplant; Haplo-Identical Transplant; Non-Myeloablative Transplant
MeSH Terms: conditions — Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Haploidentical Bone Marrow Transplant (Experimental): Participants will receive a human leucocyte antigen (HLA) haploidentical bone marrow transplantation using a non-myeloablative preparative regimen, GVHD prophylaxis.
  Interventions: Biological: Haploidentical Bone Marrow Transplantation; Biological: GVHD prophylaxis

INTERVENTIONS:
Biological: Haploidentical Bone Marrow Transplantation — The transplant preparative regimen is listed below. The - sign is the number of days before the transplant.
  * Fludarabine: 30 mg/m2 intravenously (IV) on Days -6, -5, -4, -3, and -2
  * Cyclophosphamide (Cy): 14.5 mg/kg IV on Days -6 and -5
  * Total body irradiation (TBI): 200 centigray (cGy) on Day -1
  Day 0 is the day of the infusion of non-T-cell depleted bone marrow. The bone marrow will be obtained from haploidentical related donor.
Biological: GVHD prophylaxis — The GVHD prophylaxis regimen will consist of the following:
  * Cy: 50 mg/kg IV on Days 3 and 4
  * Tacrolimus: (IV or orally) beginning on Day 5 with dose adjusted to maintain a level of 5 to 15 mg/mL
  * Mycophenolate mofetil (MMF): 15 mg/kg orally three times a day (TID) beginning on Day 5; maximum dose will be 1 g orally TID
  * Granulocyte-colony stimulating factor (G-CSF) 5 mcg/kg/day beginning on Day 5 until absolute neutrophil count (ANC) is greater than or equal to 1,000/mm^3 for 3 consecutive days

SUMMARY:
Bone marrow transplants are one treatment option for people with leukemia or lymphoma. Family members or unrelated donors with a similar type of bone marrow usually donate their bone marrow to the transplant patients. This study will evaluate the effectiveness of a new type of bone marrow transplant-one that uses lower doses of chemotherapy and bone marrow donated from family members with only partially matched bone marrow-in people with leukemia or lymphoma.

DETAILED DESCRIPTION:
Leukemia and lymphoma are types of blood cancers. Chemotherapy is a common treatment option for people with these types of cancers, but if the cancer does not respond well to chemotherapy, or if the cancer returns, a bone marrow transplant is another treatment option. In a bone marrow transplant procedure, healthy bone marrow is taken from a donor and transplanted into the patient. Bone marrow can be donated by a family member or an unrelated donor who has a similar type of bone marrow. Most bone marrow transplants are performed using a donor who is a perfect or close-to-perfect tissue match. However, for participants in this study, researchers have determined that a completely matched donor is unavailable within participants' families, and an unrelated donor match has not been found either. Participants do, however, have a family member who is a partial tissue match. Typically, people who are undergoing a bone marrow transplant receive high doses of chemotherapy before the transplant to prepare their bodies to accept the donor bone marrow. In this study, participants will undergo a new type of bone marrow transplant called a nonmyeloablative transplant, which is a reduced intensity method of transplantation that does not require high doses of chemotherapy. The purpose of the study is to examine the safety and effectiveness of a nonmyeloablative bone marrow transplant that uses partially matched bone marrow donated by a family member as a treatment option for people with leukemia or lymphoma.

This study will enroll people with leukemia or lymphoma who have a family member with a partial tissue match. Participants will be admitted to the hospital and will first receive a type of chemotherapy called fludarabine, which will be given intravenously for 5 days. In addition, another type of chemotherapy, cyclophosphamide, will be given intravenously on the first and second day. After 5 days, participants will receive a small dose of radiation. The next day, participants will undergo the bone marrow transplant. The third and fourth day after the transplant, participants will receive high doses of cyclophosphamide to help prevent two complications, graft rejection, which occurs when the body's immune system rejects the donor bone marrow, and graft-versus-host disease (GVHD), which is an attack by the donor cells on the body's normal tissues. On the fifth day after the transplant, participants will receive two additional medications, tacrolimus and mycophenolate mofetil (MMF), to help prevent GVHD; some participants may receive cyclosporine instead of tacrolimus. Participants will receive MMF for about 5 weeks and tacrolimus for about 6 months. Also beginning on the fifth day after the transplant, participants will receive daily injections of a growth factor called granulocyte-colony stimulating factor (G-CSF), which is a natural protein that increases the white blood cell count; G-CSF will be continued until a participant's white blood cell count is normal again.

Participants will remain in the hospital for approximately 2 to 3 months, but possibly longer if there are complications. While participants are in the hospital, blood samples will be collected regularly to evaluate the response and possible side effects to treatment, including GVHD. If necessary, participants will receive platelet and red blood cell transfusions. Follow-up study visits will occur 6 months and 1 year after the transplant. At Months 1, 2, 6, and 12 after the transplant, blood or bone marrow samples will be obtained. Study researchers will keep track of participants' medical condition through phone calls or mailings to participants and their doctors once a year for the rest of the participants' lives.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 21 to 70 years old; participants 1 to 21 years old are also eligible if they are ineligible for BMT CTN #0501 (NCT00412360)
* Donor must be at least 18 years of age
* Human leucocyte antigen (HLA) typing will be performed at high resolution (allele level) for the HLA-A, -B, Cw, DRB1, and -DQB1 loci. A minimum match of 5/10 is required. An unrelated donor search is not required for a person to be eligible for this study if the clinical situation dictates an urgent transplant. Clinical urgency is defined as 6 to 8 weeks from referral to transplant center or low likelihood of finding a matched, unrelated donor. The donor and recipient must be identical, as determined by high resolution typing, on at least one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA-DRB1, and HLA-DQB1. Fulfillment of this criterion shall be considered sufficient evidence that the donor and recipient share one HLA haplotype, and typing of additional family members is not required.
* Must have received cytotoxic chemotherapy within 3 months of the consent date (measured from the start date of chemotherapy)
* Acute leukemias (includes T lymphoblastic lymphoma) in the second or subsequent complete remission (CR)
* Burkitt's lymphoma in the second or subsequent CR
* Lymphoma
* Patients with adequate physical function as measured by the following:

  1. Heart: left ventricular ejection fraction at rest must be greater than or equal to 35%, or shortening fraction greater than 25%
  2. Liver: bilirubin less than or equal to 2.5 mg/dL and alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase less than five times the upper limit of normal
  3. Kidney: serum creatinine within normal range for age, or if serum creatinine is outside the normal range for age, then kidney function (creatinine clearance or glomerular filtration rate (GFR) is greater than 40 mL/min/1.73m^2
  4. Pulmonary: forced expiratory volume in one second (FEV1), forced vital capacity (FVC), and carbon monoxide diffusing capacity (DLCO) greater than 50% predicted (corrected for hemoglobin). If unable to perform pulmonary function tests, then oxygen (O2) saturation must be greater than 92% on room air.
  5. Performance status: Karnofsky/Lansky score greater than or equal to 60%

Exclusion Criteria:

* Have an HLA-matched, related, or 7 or 8/8 allele matched (HLA-A, -B, -Cw, -DRB1) related donor able to donate
* Had an autologous hematopoietic stem cell transplant in the 3 months before study entry
* Pregnant or breastfeeding
* Evidence of HIV infection or known HIV positive serology
* Current uncontrolled bacterial, viral, or fungal infection (i.e., currently taking medication with evidence of progression of clinical symptoms or radiologic findings)
* Prior allogeneic hematopoietic stem cell transplant
* History of primary idiopathic myelofibrosis

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, MS, Study Director — Center for International Blood and Marrow Transplant Research (CIBMTR), Medical College of Wisconsin
Locations (17):
- United States (17):
  - City of Hope National Medical Center, Duarte, California
  - University of California San Diego Medical Center, La Jolla, California
  - University of Florida College of Medicine (Shands), Gainesville, Florida
  - Bone Marrow Transplant Group of Georgia, Northside Hospital, Atlanta, Georgia
  - Kapi'olani Medical Center for Women and Children, University of Hawaii, Honolulu, Hawaii
  - University of Maryland, Greenbaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Comprehensive Cancer Center (SKCCC), Baltimore, Maryland
  - DFCI, Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Children's Hospital of Michigan, Detroit, Michigan
  - Washington University, Barnes Jewish Hospital, St Louis, Missouri
  - Oregon Health & Science University, Portland, Oregon
  - Fox Chase, Temple University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public.
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Result] Brunstein CG, Fuchs EJ, Carter SL, Karanes C, Costa LJ, Wu J, Devine SM, Wingard JR, Aljitawi OS, Cutler CS, Jagasia MH, Ballen KK, Eapen M, O'Donnell PV; Blood and Marrow Transplant Clinical Trials Network. Alternative donor transplantation after reduced intensity conditioning: results of parallel phase 2 trials using partially HLA-mismatched related bone marrow or unrelated double umbilical cord blood grafts. Blood. 2011 Jul 14;118(2):282-8. doi: 10.1182/blood-2011-03-344853. Epub 2011 Apr 28. PMID 21527516
- [Result] Eapen M, O'Donnell P, Brunstein CG, Wu J, Barowski K, Mendizabal A, Fuchs EJ. Mismatched related and unrelated donors for allogeneic hematopoietic cell transplantation for adults with hematologic malignancies. Biol Blood Marrow Transplant. 2014 Oct;20(10):1485-92. doi: 10.1016/j.bbmt.2014.05.015. Epub 2014 May 23. PMID 24862638

RESULTS

PARTICIPANT FLOW:
Groups:
- Haplo-marrow Transplantation: Haploidentical bone marrow transplantation using a non-myeloablative preparative regimen.
Period: Overall Study
Arm/Group | Haplo-marrow Transplantation
Started | 55
Completed | 50
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 2
Not completed — Disease Relapse/Progression | 2

BASELINE CHARACTERISTICS:
Population: Received transplant.
Arm/Group | Haplo-marrow Transplantation
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (18.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 6
  White | 40
  More than one race | 0
  Unknown or Not Reported | 1
Karnofsky Performance-status score [Number; unit: participants] — Assesses patient self-perceived global quality of life and functioning (excellent, very good, good, fair, poor), where 100 equals perfect quality of life.
  participants
    100% | 19
    90% | 19
    80% | 9
    70% | 3
Primary Disease [Number; unit: participants]
  Acute Lymphoblastic Leukemia | 6
  Acute Myelogeneous Leukemia | 22
  Biphenotypic/Undifferentiated Leukemia | 3
  Hodgkins Lymphoma | 7
  Large Cell Lymphoma | 8
  Marginal Zone B-cell Lymphoma | 1
  Mantle Cell Lymphoma | 3
Human leucocyte antigen (HLA) Typing Match Score - GVH direction [Number; unit: participants] — HLA typing will be performed at high resolution (allele level) for the HLA-A, -B, Cw, DRB1, and -DQB1 loci. A minimum match of 5/10 is required.
  participants
    5/10 | 28
    6/10 | 12
    7/10 | 9
    8/10 | 1
HLA Typing Match Score - Host vs Graft (HVG) direction [Number; unit: participants] — HLA typing will be performed at high resolution (allele level) for the HLA-A, -B, Cw, DRB1, and -DQB1 loci. A minimum match of 5/10 is required.
  participants
    5/10 | 22
    6/10 | 22
    7/10 | 3
    8/10 | 1
    9/10 | 1
    10/10 | 1
Weight [Median (Full Range); unit: kilograms] | 78 [21 to 184]

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 180 Days From the Time of Transplant
Time Frame: Measured at Month 6 and Year 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Haplo-marrow Transplantation
Number analyzed (Participants) | 50
percentage of participants
  6 months | 83.7 [70.0 to 91.5]
  1 year | 62.0 [44.1 to 75.7]

2. Secondary Outcome: Neutrophil Recovery
Description: Cumulative incidence of neutrophil recovery >500/μL at day +56
Time Frame: Measured at Days 28, 56, 90, and 100
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Haplo-marrow Transplantation
Number analyzed (Participants) | 50
percentage of participants
  Day 28 | 96.0 [89.9 to 100.0]
  Day 56 | 96.0 [89.9 to 100.0]
  Day 90 | 100.0 [96.1 to 100.0]
  Day 100 | 100.0 [96.1 to 100.0]

3. Secondary Outcome: Primary Graft Failure
Description: Primary graft failure is defined as < 5% donor chimerism on all measurements.
Time Frame: Measured at Day 67
Measure: Number; unit: participants
Arm/Group | Haplo-marrow Transplantation
Number analyzed (Participants) | 50
participants | 1

4. Secondary Outcome: Secondary Graft Failure
Description: Secondary graft failure is defined as initial recovery followed by neutropenia with < 5% donor chimerism. If no chimerism assays were performed and absolute neutrophil count is < 500/mm3, then it will be counted as a secondary graft failure.
Time Frame: Measured at Day 100
Measure: Number; unit: participants
Arm/Group | Haplo-marrow Transplantation
Number analyzed (Participants) | 50
participants | 0

5. Secondary Outcome: Platelet Recovery
Description: Platelet Recovery to 20K
Time Frame: Measured at Days 56, 90, and 100
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Haplo-marrow Transplantation
Number analyzed (Participants) | 50
percentage of participants
  Day 56 | 96.0 [89.7 to 100.0]
  Day 90 | 96.0 [89.7 to 100.0]
  Day 100 | 98.0 [93.1 to 100.0]

6. Secondary Outcome: Platelet Recovery
Description: Platelet Recovery to 50K
Time Frame: Measured at Days 56, 90, and 100
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Haplo-marrow Transplantation
Number analyzed (Participants) | 50
percentage of participants
  Day 56 | 76.0 [63.8 to 88.2]
  Day 90 | 76.0 [63.8 to 88.2]
  Day 100 | 76.0 [63.8 to 88.2]

7. Secondary Outcome: Donor Cell Engraftment
Description: Marrow or Blood Sample. Donor cell engraftment is defined as donor chimerism ≥ 5% on Day ≥ 56 after transplantation. Chimerism should be evaluated on Days ~28, ~56, ~180, and ~365 after transplantation. Chimerism may be evaluated in whole blood or mononuclear fraction.
Time Frame: Measured at Day 56
Measure: Number; unit: participants
Arm/Group | Haplo-marrow Transplantation
Number analyzed (Participants) | 50
participants
  Chimerism Performed | 42
  Donor Percentage ≥95% | 39
  Donor Percentage 5%-95% | 2
  Donor Percentage <5% | 1

8. Secondary Outcome: Acute Graft-versus-host Disease (GVHD)
Time Frame: Measured at Day 100
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Haplo-marrow Transplantation
Number analyzed (Participants) | 50
percentage of participants
  Grade II-IV Acute GVHD | 32.0 [18.9 to 45.1]
  Grade III-IV Acute GVHD | 0.0 [0.0 to 0.0]

9. Secondary Outcome: Chronic GVHD
Time Frame: Measured at Year 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Haplo-marrow Transplantation
Number analyzed (Participants) | 50
percentage of participants | 12.9 [2.9 to 22.9]

10. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the minimum time interval of the times to relapse/recurrence, to death or to last follow-up.
Time Frame: Measured at Year 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Haplo-marrow Transplantation
Number analyzed (Participants) | 50
percentage of participants | 47.9 [32.0 to 62.2]

11. Secondary Outcome: Treatment-related Mortality (TRM)
Time Frame: Measured at 6 months and 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Haplo-marrow Transplantation
Number analyzed (Participants) | 50
percentage of participants
  6 months | 4.0 [0.0 to 9.5]
  1 year | 7.0 [0.0 to 15.0]

12. Secondary Outcome: Infections
Description: Number of infections; infections will be reported by anatomic site, date of onset, organism and resolution, if any. Patients will be followed for infection for 1 year post-transplant.
Time Frame: Measured at Year 1
Population: 36 patients incurred a total number of 108 infection events.
Measure: Number; unit: participants
Arm/Group | Haplo-marrow Transplantation
Number analyzed (Participants) | 50
participants
  1 Infection | 14
  2 Infections | 6
  3 Infections | 10
  4 Infections | 2
  5 Infections | 1
  6-10 Infections | 2
  >10 Infections | 1

ADVERSE EVENTS:
Time Frame: 1-year post-transplant
Description: Serious adverse events are defined as events associated with death, life-threatening event, disability, congenital anomaly, required intervention to prevent permanent impairment or damage, hospitalization or other serious adverse event.
Arm/Group | Haplo-marrow Transplantation
Serious Adverse Events (participants affected / at risk) | 5/52
Other Adverse Events (participants affected / at risk) | 1/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haplo-marrow Transplantation (N=52)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.92% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haplo-marrow Transplantation (N=52)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2009-01-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT00849147/Prot_SAP_ICF_000.pdf